CLINICAL TRIAL: NCT03055793
Title: A Real Life, on International, Multicenter Study to Assess the Efficacy and Quality of Life in Greek Asthmatic Patients Who Will be on Fixed Dose Bodesonide Formoterol Combination Treatment
Brief Title: Quality of Life Assessment in Greek asthmatIc Patients Treated With the Fixed Dose Combination of Budesonide / Formoterol in Clinical Practice
Acronym: SKIRON
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-HAL-EL-70
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Asthma; Quality of Life; Satisfaction
MeSH Terms: conditions — Asthma; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: budesonide formoterol fixed combination — Asthmatic patients who will be on budesonide formoterol fixed combination treatment administered by Elpenhaler device.

SUMMARY:
The greater efficacy of combination therapy led to the development of fixed combination devices which simultaneously carry both glucocorticosteroid and a LABA (eg stable combinations of fluticasone-salmeterol, budesonide-formoterol).

Fixed combinations are easier to use for patients, potentially increasing compliance, and ensure that the LABA always accompanied by glycocorticosteroeides1. From the available combinations of the combination of budesonide-formoterol can be used both in maintenance therapy and for the relief of symptoms due to the rapid onset of action of formoterol compared with salmeterol. Both components of budesonide-formoterol combination when administered on demand contribute to strengthening protection from severe exacerbations in patients receiving combination therapy for maintenance, and enable improvement of asthma control at relatively low doses of ICS.

DETAILED DESCRIPTION:
This prospective observational study of the Greek population to approximately 2,500 patients suffering from asthma, aims to collect the characteristics of patients that were selected to obtain an inhaled combination of budesonide and formoterol fumarate dihydrate in any of portions 100 / 6mcg, 200 / 6mcg, 400/12 mcg (Pulmoton®), and to collect data on the quality of life to such an inhaled combination through Elpenhaler® device.

Data will be collected for a period of three months from patients diagnosed with asthma not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting or patients already adequately controlled on both inhaled corticosteroids and long-acting beta2-agonists.

Data will be collected during the period of one (1) to three (3) months (± 2 weeks) from the initiation of treatment with inhaled combination include ACQ checklist questionnaire mini AQLQ, questionnaire FSI 10, and data any existing comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Men or women patients with asthma over 18 years
* Compliant to treatment
* Compliant to the study procedures
* Signed consent form after written study information
* Patients with Asthma to start treatment with the inhaled combination of budesonide / formoterol at doses 100 / 6mcg, 200 / 6mcg, 400/12 mcg, through Elpenhaler® device may be included in the study. Under current SPC, the drug Pulmoton® indicated in the regular treatment of asthma, wherein the administration of the combination (inhaled corticosteroid and long-action beta2-agonist) is appropriate, namely in patients:
* patients not adequately controlled with inhaled corticosteroids and 'as needed' inhaled beta2-agonists short-acting or
* already adequately controlled on both inhaled corticosteroids and long-acting beta2-agonists Note: Pulmoton® 100/6 micrograms / dose is not suitable for patients with severe asthma.

Exclusion Criteria:

* Men or women with Asthma patients under 18 years
* Non-compliance to treatment
* Non-compliance to study procedures
* Do not signed patient consent
* Incorrect use of inhaled therapies
* Patients with COPD (any stage)
* Patients already receiving any combination ICS / LABA at entry into the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Efficacy (ACQ score) | 3 months
  ACQ score

SECONDARY OUTCOMES:
Quality of Life (AQLQ score) | 3 months
  AQLQ score
Patient Satisfaction (FS1 -10 score) | 3 months
  FS1 -10 score

CONTACTS AND LOCATIONS:
Locations (1):
- 7th Pulmonary Dept, Athens Chest Hospital, Athens, Mesogion Ave. 152, Greece

IPD SHARING:
Plan to Share IPD: No